CLINICAL TRIAL: NCT00755508
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Multicenter, Proof-of-Concept Study to Evaluate the Safety and Efficacy of ROZEREM™ Taken in Combination With Gabapentin for the Treatment of Subjects With Chronic Insomnia
Brief Title: Efficacy and Safety of Ramelteon Combined With Gabapentin in Treating Patients With Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-05-TL-375-055; U1111-1114-3348 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Chronic Insomnia; DIMS (Disorders of Initiating and Maintaining Sleep); Disorders of Initiating and Maintaining Sleep; Insomnia Disorder Sleep Initiation Dysfunction; Transient Insomnia; Drug Therapy; Sleep Disorders, Intrinsic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Disorders, Intrinsic | interventions — ramelteon; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Ramelteon 4 mg QD and Gabapentin 400 mg QD (Experimental)
  Interventions: Drug: Ramelteon and gabapentin
- Ramelteon 8 mg QD and Gabapentin 800 mg QD (Experimental)
  Interventions: Drug: Ramelteon and gabapentin
- Ramelteon 8 mg QD and Gabapentin Placebo QD (Experimental)
  Interventions: Drug: Ramelteon
- Gabapentin 800 mg QD (Active Comparator)
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon and gabapentin — Ramelteon 4 mg, tablets, orally, once daily and gabapentin 400 mg, capsules, orally, once daily for up to one week.
  Other Names: TAK-375; Ramelteon; Neurontin®; Rozerem
  Arms: Ramelteon 4 mg QD and Gabapentin 400 mg QD
Drug: Ramelteon and gabapentin — Ramelteon 8 mg, tablets, orally, once daily and gabapentin 800 mg, capsules, orally, once daily for up to one week.
  Other Names: TAK-375; Ramelteon; Neurontin®; Rozerem
  Arms: Ramelteon 8 mg QD and Gabapentin 800 mg QD
Drug: Ramelteon — Ramelteon 8 mg, tablets, orally, once daily and gabapentin placebo-matching capsules, orally, once daily for up to one week.
  Other Names: TAK-375; Rozerem
  Arms: Ramelteon 8 mg QD and Gabapentin Placebo QD
Drug: Gabapentin — Ramelteon placebo-matching tablets, orally, once daily and gabapentin 800 mg, capsules, orally, once daily for up to one week.
  Other Names: Neurontin®; Rozerem
  Arms: Gabapentin 800 mg QD
Drug: Placebo — Ramelteon placebo-matching tablets, orally, once daily and gabapentin placebo-matching capsules, orally, once daily for up to one week.
  Other Names: Rozerem
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of ramelteon, once daily (QD), taken in combination with Gabapentin for treating insomnia.

DETAILED DESCRIPTION:
Approximately 60 to 70 million adults in the United States alone are affected by insomnia. Daytime symptoms of insomnia include tiredness, lack of energy, difficulty concentrating, and irritability. Recent epidemiologic research focusing on quality of life has identified significant insomnia-related morbidities that relate to work productivity, health care utilization, and risk of depression. Insomnia is also associated with diminished work output, absenteeism, and greater rates of accidents. gamma-aminobutyric acid is the major inhibitory transmitter in the central nervous system and most currently prescribed sleep agents are benzodiazepine receptor agonists, which induce sleep by binding to the benzodiazepine receptor site of the gamma-aminobutyric acid -A receptor complex. In addition to sleep, benzodiazepine receptor agonists can cause a wide range of ancillary effects not directly related to sleep, including sedative, anxiolytic, muscle-relaxant, and amnesic effects, and have risks of tolerance, dependence, and abuse potential.

Gabapentin is a novel anti-epileptic drug, which is currently used in subjects with partial seizures. Some studies have shown that gabapentin also has an effect on sleep architecture. In several studies, which included healthy subjects, epileptic subjects, and subjects with restless leg syndrome, the use of gabapentin been shown to prolong slow-wave sleep, increase total sleep time and sleep efficiency, and decrease number of awakenings.

Ramelteon is a melatonin receptor agonist with affinity for the human melatonin receptor subtype 1, melatonin receptor subtype 2 and selectivity over the melatonin receptor subtype 3 receptor. It also demonstrates agonist activity in vitro relative to melatonin in cells expressing human melatonin receptor subtype 1 or melatonin receptor subtype 2 receptors. The binding of melatonin at these receptors is thought to contribute to maintenance of the circadian rhythm underlying the normal sleep-wake cycle.

The purpose of this trial is to determine if the co-administration of Ramelteon and gabapentin may produce increased sleep efficiency through reduction of wake time after persistent sleep onset, in addition to the reduction in sleep latency and increase in sleep duration. Study participation is anticipated to be about one month.

ELIGIBILITY:
Inclusion Criteria:

* Female patients of childbearing potential must be nonpregnant and nonlactating, and utilizing an acceptable method of contraception.
* Based on sleep history, the subject has had primary insomnia as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised (DSM-IV-TR™) for at least 3 months.
* Based on sleep history, reports a subjective sleep latency greater than or equal to 45 minutes and reports wake time after persistent sleep onset of greater than or equal to 45 minutes.
* Has an average wake time after persistent sleep onset of at least 60 minutes as determined by polysomnography during Screening (Day minus 7 PM through Day minus 5 AM). Wake time after persistent sleep onset must be greater than or equal to 30 minutes each night of polysomnography Screening.
* Reports wake time after persistent sleep onset values of at least 60 minutes on at least 3 of the 7 nights during the single-blind screening period (Day minus 6 AM through Day 1 AM) as determined by post-sleep questionnaire.
* Has an average latency to persistent sleep of at least 20 minutes as determined by polysomnography during Screening (Day minus 7 PM through Day minus 5 AM).
* Based on sleep history, has an habitual bedtime between 9:00 PM and 1:00 AM.
* The subject is willing to have a fixed bedtime and agrees to go to bed within plus or minus 30 minutes of the habitual bedtime during the entire study and agrees to remain in bed for at least 8 hours each night.
* Based on sleep history, has not been using pharmacological assistance to sleep or uses pharmacological assistance no more than 4 times per week during the 3 months prior to Initial Screening.
* Has consistent access to a touch-tone phone and are willing to complete telephone questionnaires twice daily during participation in the study.

Exclusion Criteria:

* Has a known hypersensitivity to gabapentin or its ingredients, ramelteon or related compounds, including melatonin, and 5-hydroxytryptophan.
* Has participated in any other investigational study and/or taken any investigational drug within 30 days prior to the first dose of single-blind study medication.
* Has sleep schedule changes required by employment (eg, shift worker) within 3 months prior to the first dose of single-blind study medication.
* Has flown across greater than 3 time zones within 7 days prior to Initial Screening, or will travel across 2 or more time zones during the course of the study.
* Has participated in a weight loss program or has substantially altered their exercise routine within 30 days prior to the first dose of single-blind study medication.
* Has ever had a history of seizures, sleep apnea, and/or chronic obstructive pulmonary disease.
* Has a history of psychiatric disorder (including anxiety, depression, mental retardation, cognitive disorder, bipolar illness and schizophrenia) within the past 6 months of Initial Screening.
* Has a history of fibromyalgia.
* Has a history of drug addiction or drug abuse within the past 12 months of Initial Screening.
* Has a history of alcohol abuse within the past 12 months, as defined in DSM-IV-TR™ and/or regularly consumes more than 2 alcoholic drinks per day.
* Has a current significant hepatic, endocrine, cardiovascular, gastrointestinal, pulmonary, hematological, metabolic or neurological disorders, unless currently controlled and stable with protocol-allowed medication, within 30 days prior to the first dose of single-blind study medication.
* Has any diagnosed renal impairment within 30 days prior to the first dose of single-blind study medication.
* Has a previous history of cancer, other than basal cell carcinoma, that has not been in remission for at least 5 years prior to the first dose of single-blind study drug.
* Uses tobacco products or any other products that may interfere with the sleep wake cycle during nightly awakenings.
* Is required to take or intends to continue taking any disallowed medication or any prescription medication or over-the counter medication that is known to affect the sleep/wake function or otherwise interfere with evaluation of the study medication, including:

  * Anxiolytics central nervous system active drugs (including herbal)
  * Hypnotics Narcotic analgesics
  * Antidepressants Beta blockers
  * Anticonvulsants St. John's Wort
  * Sedating H1 antihistamines Kava-kava
  * Systemic steroids Ginkgo-biloba
  * Respiratory stimulants over-the counter and prescription stimulants
  * Sedating decongestants over-the counter and prescription diet aids
  * Antipsychotics over-the counter sleep aids
  * Muscle relaxants Antacids
  * Melatonin and all other drugs or supplements known to affect sleep/wake function.
* Has a positive hepatitis panel including anti- hepatitis A virus, hepatitis B surface antigen or anti-hepatitis C virus.
* Has a positive urine drug screen including alcohol at Initial Screening or a positive breathalyzer test at each polysomnography Screening check-in.
* Has an apnea hypopnea index (per hour of sleep) >15 as seen on polysomnography, on the first night of the polysomnography screening.
* Has a history of restless leg syndrome.
* The subject has a body mass index of less than 18 or greater than 34 (weight /height2).
* Has any additional condition(s) that in the Investigator's opinion would:

  * Affect sleep/wake function
  * Prohibit the subject from completing the study
  * Not be in the best interest of the subject.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2005-11; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Mean objective wake time after persistent sleep onset in sleep lab. | Nights: 1 and 2.

SECONDARY OUTCOMES:
Subjective wake time after persistent sleep onset determined by the post-sleep questionnaire. | Nights: 1, 2, 3, 4, 5, 6 and 7.
Number of awakenings after persistent sleep polysomnography. | Nights: 1 and 2
Subjective number of awakenings as determined by post-sleep questionnaire. | Nights: 1, 2, 3, 4, 5, 6 and 7.
Latency to persistent sleep and total sleep time as determined by polysomnography. | Nights: 1 and 2
Subjective sleep latency, subjective total sleep time and subjective sleep quality determined by post-sleep questionnaire. | Nights: 1, 2, 3, 4, 5, 6 and 7.
Daytime functioning determined by pre-sleep questionnaire. | Nights: 1, 2, 3, 4, 5, 6 and 7.

CONTACTS AND LOCATIONS:
Overall Officials: Sr. VP Clinical Science, Study Director — Takeda

REFERENCES:
- See also: Rozerem Package Insert. — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI